CLINICAL TRIAL: NCT01097837
Title: Epilepsy Birth Control Registry
Acronym: EBCR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuroendocrine Associates P.C. (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Andrew G. Herzog M.D., M.Sc., Principal Investigator, Neuroendocrine Associates P.C.
Other Study IDs: 137557
Record Dates: First submitted 2010-03-31; First posted 2010-04-02 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Epilepsy
Keywords: Epilepsy; Contraceptive; Birth Control; Seizure; This study is looking at the use of different birth control measures in women with epilepsy.
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Epilepsy: Cohort is comprised of women with epilepsy between 18 and 47.
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — This is an observational study conducted by anonymous survey. There is no intervention.

SUMMARY:
Despite the importance of birth control to women of reproductive age, there has been little formal investigation of the safety and effectiveness of birth control methods in women with epilepsy. To remedy this, doctors from Harvard and Columbia University Medical Schools have developed a website that offers a survey to help us gain more knowledge and some educational material that will be updated regularly to provide the latest information. The ultimate goal is to develop guidelines for the selection of safe and effective birth control methods and to make sure that the best forms of birth control become available to women with epilepsy in all communities of our society.

Go to www.epilepsybirthcontrolregistry.com take our survey and then catch up on the latest information about birth control for women with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Women with Epilepsy between 18 and 47

Exclusion Criteria:

* Women without epilepsy
* Women under 18
* Women over 47

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants are women with epilepsy between the ages of 18 and 47.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-03; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of seizures on hormonal versus non-hormonal contraception, stratified by antiepileptic drug category | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrew G Herzog, M.D.,M.Sc., Principal Investigator — Neuroendocrine Associates P.C.
Locations (2):
- United States (2):
  - Neuroendocrine Associates P.C., Wellesley, Massachusetts
  - Columbia University Medical Center, New York, New York